CLINICAL TRIAL: NCT06197763
Title: Impact of Therapy Using Colesevelam Treatment Reducing Bile Acids in Patients With Fontan Circulation (MYSTIC) Pilot Study.
Brief Title: Impact of Therapy Using Colesevelam Treatment Reducing Bile Acids in Patients With Fontan Circulation.
Acronym: MYSTIC
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: St. Boniface Hospital (Other)
Responsible Party: Principal Investigator, Dr. Ashish Shah, Qualified Investigator, St. Boniface Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CTA/2023/001
Record Dates: First submitted 2023-10-04; First posted 2024-01-09 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Fontan Circulation
MeSH Terms: interventions — Colesevelam Hydrochloride

STUDY DESIGN:
Intervention Model Description: prospective, double-blind, placebo cross-over, pilot study evaluating colesevelam (intestinal BA scavenger) therapy and placebo in 25 stable adult FC participants. These participants will be recruited from the cardiology clinics at the St. Boniface Hospital, specifically the Manitoba Adult Congenital Heart (MACH) Clinic.
  A further 25 age- and sex- matched healthy control participants will be recruited from advertising at St. Boniface Hospital and University of Manitoba. Healthy controls will only undergo the baseline visit and will not receive the investigational drug or placebo.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants, investigators, and everyone involved in study conduct or analysis or with any other interest in this double-blind study will remain blinded with regard to the randomization treatment assignments until after data collection completion. The access to the randomization code will be kept restricted until its release for analysis.
  The DSMB will be provided with unblinded data in order to allow them to review efficacy and safety and to fulfill their tasks as outlined in the DSMB charter.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Fontan participants (Experimental): Participants will be randomized to be treated with either colesevelam (625 mg tablets - 3 tables twice per day) or placebo (3 tablets twice per day) for 6 weeks, interspersed by 8 week of washout time.
  Interventions: Drug: Colesevelam
- Healthy control participants (Sham Comparator): These healthy control participants will be comparators to the randomized Fontan participants. Healthy controls will only undergo the baseline visit and will not receive the investigational drug or placebo.
  Interventions: Other: Control Arm

INTERVENTIONS:
Drug: Colesevelam — 625 mg tablets - 3 tables twice per day of Colesevelam or placebo for 6 weeks (crossover), interspersed by 8 week of washout time.
  Arms: Fontan participants
Other: Control Arm — No Treatment: baseline assessment only
  Arms: Healthy control participants

SUMMARY:
This is the first pilot study proposing a novel therapeutic option treating patients with Fontan circulation (FC), a high-risk condition that has no definite treatment options available, other than heart or heart-liver transplantation. The investigator's identification of elevated BA and their association with adverse clinical - investigational features in Fontan patients are novel.

DETAILED DESCRIPTION:
The investigators propose a prospective, double-blind, placebo cross-over, pilot study evaluating colesevelam (intestinal BA scavenger) therapy and placebo in 25 stable adult FC participants. These participants will be recruited from the cardiology clinics at the St. Boniface Hospital, specifically the Manitoba Adult Congenital Heart (MACH) Clinic. Participants will be randomized to be treated with either colesevelam (625 mg tablets - 3 tables twice per day) or placebo (3 tablets twice per day) for 6 weeks, interspersed by 8 week of washout time. Local research and ethics board approval will be obtained. Informed consent will be obtained from all participants.

A further 25 age- and sex- matched healthy control participants will be recruited from advertising at St. Boniface Hospital and University of Manitoba. These healthy control participants will be comparators to the randomized Fontan participants at baseline. Recruitment of this group will be completed after all Fontan participants have been screened, consented, and randomized to ensure accuracy of age and sex matching. Age and sex matched participants will be +/- 3 years and not pregnant or nursing at time of study visit.

ELIGIBILITY:
Inclusion criteria - Fontan participants

i) Of full age of consent (at least ≥ 18 years of age) at screening

ii) Signed and dated written informed consent in accordance with ICF-GCP and local regulations prior to admission to the study

iii) Male or female participants. Women of childbearing potential (WOCBP) must be ready and able to use highly effective methods of birth control that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in the participant informed consent form.

iv) Diagnosis of Fontan circulation documented in the participant's medical record

Inclusion criteria - Healthy control participants

i) Of full age of consent (at least ≥ 18 years of age) at screening

ii) Signed and dated written informed consent in accordance with ICF-GCP and local regulations prior to admission to the study

iii) Male or female participants

Exclusion criteria - Fontan participants

i) Has previously received a heart or heart-liver transplant

ii) Contraindication for using colesevelam, including allergy

iii) Any physical or mental condition significantly affecting the participant's ability to participate in the investigator's opinion

iv) Women who are pregnant, nursing, or who plan to become pregnant while in the trial

Exclusion criteria - Healthy control participants

i) Any known medical condition

ii) Any physical or mental condition significantly affecting the participant's ability to participate in the investigator's opinion

iii) Women who are pregnant or nursing at time of study visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Drug safety | 20 Weeks
  This outcome will be evaluated by identifying side effects experienced by any of the study participants throughout the study period.
  This information will be collected during biweekly phone calls to each of the study participants by the study coordinator. The study participants will also have the contact number of the study coordinator to notify them of any issues.
  The investigators have also established a "Data and drug safety monitoring board" which will review each of the side effects experienced by the study participants.
Drug compliance | 20 weeks
  This will be evaluated by checking with each study participant about their drug compliance and identifying the number of days, they have taken tablets as recommended.
Impact of colesevelam on plasma & stool bile acid concentration. | 20 Weeks
  Plasma & stool bile acid concentration (total and their subcomponents) will be measured at baseline as well as after medication (placebo & colesevelam) use.

SECONDARY OUTCOMES:
Impact of colesevelam on blood & urine metabolites. | 20 Weeks
  Plasma and urine metabolites will be measured before and after the drug (colesevelam) and placebo therapy.
Impact of colesevelam on gut microbiome. | 20 Weeks
  Stool samples before and after each medication (placebo and colesevelam) use will be analyzed to determine gut microbiome composition at baseline, and the impact of the colesevelam therapy on this composition.
Impact of colesevelam on hemodynamics. | 20 Weeks
  Each study participant will be evaluated by total body-impedance-based, non-invasive cardiac system (NICaS) derived hemodynamic parameters (cardiac output, cardiac index, stroke volume, stroke index, cardiac power output), before and after medication (placebo & colesevelam) use.
Gut microbiome comparison between healthy subjects and Fontan patients. | Baseline
  The gut microbiome will be compared between healthy subjects and patients with Fontan circulation at baseline.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shah AH, Armstrong HK, Mittal I, Reimer A, Kunutsor SK, Ducas RA, Alizadeh K, Tam JW, Ravandi A, Dhingra S. IMpact of therapY using coleSevelam treatment reducing bile acids in patients with fonTan cIrCulation (MYSTIC): Rationale and study design. Am Heart J. 2026 Jan;291:81-88. doi: 10.1016/j.ahj.2025.08.011. Epub 2025 Aug 19. PMID 40840821